CLINICAL TRIAL: NCT07054723
Title: Daily Stress Process and Daily Cognitive Performance Among Racially Diverse Breast Cancer Survivors: A Feasibility and Validation Study
Brief Title: Surviving Daily Life
Acronym: GOCE
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: iRISID-2025-0027; JT 44399 (Other: JeffTrial Number)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Stress; Cognitive Change; Breast Cancer; Breast Carcinoma; Breast Neoplasm; Cognitive Dysfunction
Keywords: Mobile Survey; Daily Diary; Breast Cancer Survivors
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mobile Daily Diary Survey: Participants in the study will be given a mobile phone to complete the study. Participants will first complete the baseline survey using the mobile phone (day 1) to collect demographic and socioeconomic status information. Starting from day 2 to day 14, participants will complete the short morning (2-3 min) and slightly longer (5-7 min) evening mobile daily diary surveys. The morning survey asks questions about sleep, morning outlook, and anticipatory stress and positive experiences. The evening survey asks questions about the respondent's daily experiences (stressors, mood, physical symptoms). After each survey, respondents will complete three brief objective cognitive tasks. To minimize the risk of data breach, all the information from the survey will be stored on a password protected mobile phone which will be set up to ensure that participants are only able to use the phone for the study processes, not for phone calls or to connect to the internet.
  Interventions: Behavioral: Mobile Daily Diary

INTERVENTIONS:
Behavioral: Mobile Daily Diary — This study will include a 14-day daily diary survey in which participants will be expected to complete morning (~5 minutes) and night (~10 minutes) assessments using mobile phones provided by the research team.

SUMMARY:
The primary goal of this project is to evaluate the feasibility of a 14-day mobile daily diary study among racially diverse breast cancer survivors. Further, the investigators will examine the validity and reliability of the daily stress and daily cognitive performance measures among breast cancer survivors. This pilot project will recruit 30 racially diverse breast cancer survivors (Asian, Black, Latina, and white; ages 40 and older; at least five years post-diagnosis) who are patients at the Sidney Kimmel Comprehensive Cancer Center. The daily diary survey questions will be available in English, Spanish, and Chinese to accommodate the preferred language of the target participants.

DETAILED DESCRIPTION:
This is a pilot study that will assess the feasibility of a 14-day mobile daily diary survey to measure daily stress and cognitive performance among long-term breast cancer survivors.

Participants will be recruited from the Sidney Kimmel Cancer Center (SKCC) at Thomas Jefferson University (TJU). Potential participants will be identified via the SKCC/TJU Tumor Registry. Potential participants will be contacted with their cancer care team approval. Contact may be accomplished via an upcoming clinical appointment, phone, email, or MyChart (RLS) depending on the patient's communication preference or clinical team guidance.

Participants will start study procedures by completing the baseline survey using the mobile phone (day 1) to collect demographic and socioeconomic status information. Starting from day 2 to day 14, participants will complete the short morning (2-3 min) and slightly longer (5-7 min) evening mobile daily diary surveys. The morning survey asks questions about sleep, morning outlook, and anticipatory stress and positive experiences. The evening survey asks questions about the respondent's daily experiences (stressors, mood, physical symptoms). After each survey, respondents will complete three brief objective cognitive tasks. To minimize the risk of data breach, all the information from the survey will be stored on the password protected study mobile phone. The study mobile phones will be set up to ensure that it can only be used for study purposes, that is, participants are unable to make phone calls or connect to the internet with the study phone.

Findings from this pilot project will provide critical preliminary evidence regarding the feasibility of a mobile daily diary method among racially diverse breast cancer survivors, as well as the reliability and validity of the important measures related to daily stress, daily cognitive performance, and daily cognitive problems in racially diverse populations.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study:

* Individuals 40 or older
* Five or more years after breast cancer diagnosis
* Self-identified as Asian, Black, Latina, or white
* Able to read in English, Spanish, or Chinese

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Under 40
* Cannot provide informed consent

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivor who self-identifies as White, Black/African American, Latina, or Asian
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Completion rate of the 14-day mobile daily diary survey | Daily, from Day 2 through Day 15
  The feasibility of the mobile daily diary method will be based on calculating the percentage of completed daily diary surveys as well as percentages of completed morning and evening surveys. An accepted completion rate is predetermined at the level of 70% or higher

SECONDARY OUTCOMES:
predictive validity of the Daily Inventory of Stressful Experiences (DISE) | Daily, from Day 2 through Day 15
  Predictive validity of the daily stressor exposure and severity will be conducted by testing the within-person and between-person associations between daily stressor exposure and severity with daily negative and positive affect, daily cognitive performance, and daily cognitive problems.
predictive validity of Ambulatory Cognitive Assessment measures | Twice Daily, from Day 2 through Day 15
  Construct validity of the daily cognitive assessment measures will be assessed by conducting a multilevel confirmatory factor analysis (CFA) to assess the fit of our hypothesized measurement model.
internal reliability of Ambulatory Cognitive Assessment measures | Twice Daily, from Day 2 through Day 15
  Between-person reliability (higher intraclass correlation is expected, thus no calculation of within-person reliability) by calculating internal consistency (i.e., Cronbach's alpha) across all persons and days.
internal reliability of Cognitive Interference and Memory Lapses scale | Daily, from Day 2 through Day 15
  Between-person reliability (higher intraclass correlation is expected, thus no calculation of within-person reliability) by calculating internal consistency (i.e., Cronbach's alpha) across all persons and days.
  PROMIS® v2.0 - Cognitive Function
  Scoring:
  * Raw Score Range: Varies by short form:
  * 4-item: 4-20
  * 6-item: 6-30
  * 8-item: 8-40 T-Score Range: ~22 to 65
  * Mean: 50
  * Standard Deviation: 10
  Interpretation:
  * Higher scores indicate better cognitive function (i.e., less cognitive interference).
  * A T-score of 60 means one SD above average (better functioning); a T-score of 40 means one SD below average (more interference)
  Montreal Cognitive Assessment (MoCA)
  Scoring:
  * Total Score Range: 0-30
  * Cutoff for Normal Cognition: ≥26
  Interpretation:
  * Higher scores indicate better memory and cognitive function.
  * Scores between 22-25 suggest mild cognitive impairment (MCI).
  * Scores below 22 may indicate more significant memory or cognitive issues

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Lopez, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No